CLINICAL TRIAL: NCT06851559
Title: A Phase 2, Randomized, Double-Blind, Multi-Center Study in Adult Subjects With Eosinophilic Esophagitis (EoE) to Evaluate the Safety and Efficacy of Vonoprazan 20 mg Compared to Placebo After 12 Weeks and to Evaluate the Safety and Efficacy of Vonoprazan 20 mg Up to 24 Weeks
Brief Title: A Study in Adult Participants With EoE to Evaluate Vonoprazan 20 mg Compared to Placebo After 12 Weeks and to Evaluate Vonoprazan 20 mg Up to 24 Weeks
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EoE-201
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: Vonoprazan; Adults
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Intervention Model Description: The study will enroll participants ≥18 years of age.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vonoprazan 20 mg (Experimental): Participants will be administered vonoprazan at a dose of 20 mg for 12 weeks. Participants will continue to receive the same dose for an additional 12 weeks.
  Interventions: Drug: Vonoprazan
- Placebo (Experimental): Participants will be administered placebo for 12 weeks. Participants will then receive vonoprazan 20 mg for an additional 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan will be administered orally as a tablet
  Arms: Vonoprazan 20 mg
Drug: Placebo — Placebo will be administered orally as tablet
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of vonoprazan 20 mg once daily (QD) compared to placebo QD in the number of participants with a peak eosinophilic histologic response <15 eosinophils per high-power field (eos/hpf) after 12 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* The participant is ≥18 years of age at the time of informed consent signing.
* In the opinion of the investigator or subinvestigators, the participant is capable of understanding and complying with protocol requirements, including completion and compliance with the electronic diary. The diary must be completed on at least 11 of the last 14 days in the 2 weeks prior to Visit 2 (Day -1).
* The participant signs and dates a written informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures.
* The participant has a peak eosinophil count of at least 15 eos/hpf [X 400] from at least 2 of the 3 esophageal levels on screening endoscopy as measured in at least 6 biopsies, at least 2 each from the proximal, mid, and distal segments of the esophagus based on central reading.
* The participant has 4 or more days with dysphagia episodes documented via electronic diary in the 2 weeks prior to Visit 2 (Day -1).
* The participant must remain on a stable diet for at least 6 weeks prior to the Screening Period and is expected to remain on a stable diet during the course of the study; stable diet is defined as not initiating new elimination diets or reintroducing previously eliminated foods.
* A female participant of childbearing potential who is or may be sexually active with a non-sterilized male partner agrees to routinely use adequate contraception from the signing of informed consent until 4 weeks after the last dose of study drug.

Exclusion Criteria:

* The participant is on a pure liquid diet.
* The participant has documented erosive esophagitis at the screening endoscopy.
* The participant has other known causes of esophageal eosinophilia or either of the following conditions: hypereosinophilic syndrome, or eosinophilic granulomatosis with polyangiitis (Churg-Strauss Syndrome).
* The participant has a documented diagnosis of eosinophilic gastritis, duodenitis, jejunitis, ileitis, proctitis, or colitis.
* The participant has endoscopic Barrett's esophagus (>1 cm of columnar-lined esophagus) or dysplastic changes in the esophagus.
* The participant has a history of achalasia, Crohn's disease, ulcerative colitis, or celiac disease.
* The participant has a known active Helicobacter pylori infection.
* The participant has any other clinically significant structural conditions affecting the esophagus, including: esophageal varices, viral or fungal infection, and history of radiation therapy, radiofrequency ablation, endoscopic mucosal resection, cryotherapy to the esophagus, caustic or physiochemical trauma (including sclerotherapy or esophageal variceal band ligation), or esophageal surgery.
* The participant has a history of surgery or non-EoE endoscopic intervention, such as gastric bypass, fundoplication, gastric sleeve, or a history of gastric or duodenal surgery (except endoscopic removal of benign polyps).
* The participant has gastric ulcer(s) or duodenal ulcer(s) within 4 weeks before the first dose of study drug.
* The participant has had clinically significant upper or lower gastrointestinal bleeding within 4 weeks prior to the Screening Period.
* The participant has esophageal stricture(s) unable to be passed with an 8 to 10 mm endoscope, clinically requires dilation, or has a history of dilation within the 3 months prior to the Screening Period.
* Use of prescription or non-prescription PPIs or PCABs within 2 months prior to the Screening Period.
* Use of swallowed topical corticosteroid or budesonide oral suspension for EoE within 2 months prior to the Screening Period.
* Use of systemic corticosteroid for any condition within 3 months prior to the Screening Period.
* Use of inhaled or nasal glucocorticoids within 3 months prior to the Screening Period, except stable dose for at least 3 months prior to the Screening Period for any condition (should not be changed during the study).
* Use of dupilumab within 3 months prior to the Screening Period.
* The participant has received any investigational compound within 30 days or any investigational biologic within 3 months prior to the start of the Screening Period (including those in post-marketing studies) or vonoprazan in a clinical trial at any time. A participant who has been screen failed from another clinical study and who has not been dosed may be considered for enrollment in this study.
* The participant has used immunomodulatory therapy within 3 months prior to the Screening Period or anticipates using immunomodulatory therapy during the study (except for any ongoing regimen of allergy therapy).
* The participant is a study site employee, an immediate family member, is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling), or who may have consented under duress.
* The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, ascorbic acid, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, titanium oxide, or red ferric oxide). Skin testing may be performed according to local standard practice to confirm hypersensitivity.
* The participant has a history of alcohol abuse, illegal drug use, drug addiction or regularly consumes alcohol within the 12 months prior to the Screening Period (based on self-report). Participants must have a negative urine drug screen for non-prescribed medications at screening. Participants taking prescription drugs will be allowed. Occasional, recreational use of cannabis is allowed. However, participants with a cannabis use disorder (eg, frequent use, functional-social impairment, withdrawal symptoms) per the opinion of the investigator should be excluded.
* The participant is taking any excluded medications or treatments listed in the protocol.
* If female, the participant is pregnant, lactating, or intending to become pregnant before, during, or within 4 weeks after participating in this study, or intending to donate ova during such time period.
* The participant has a history or clinical manifestations of significant central nervous system, cardiovascular, pulmonary, metabolic, other gastrointestinal, urological, endocrine, or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participant safety.
* The participant has a history of malignancy (including MALToma) or has been treated for malignancy within 5 years prior to the start of the Screening Period (Visit 1). The participant may be included in the study if he/she has recovered from cutaneous basal cell carcinoma or cervical carcinoma in situ.
* The participant has acquired immunodeficiency syndrome or human immunodeficiency virus infection, or tests positive for the hepatitis B surface antigen, hepatitis C virus (HCV) antibody, or HCV-ribonucleic acid (RNA). However, participants who test positive for HCV antibody but negative for HCV-RNA are permitted to participate.
* The participant has Zollinger-Ellison syndrome or other gastric acid hypersecretory conditions.
* The participant requires hospitalization or has surgery scheduled during the course of the study or has undergone major surgical procedures within 30 days prior to the Screening Period.
* The participant has moderate to severe hepatic impairment (Child-Pugh Class B and Child-Pugh Class C).
* The participant has severe renal impairment (estimated glomerular filtration rate <30 mL/min).
* The participant has any of the following abnormal laboratory test values at the start of the Screening Period:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >2 × ULN (except participants with Gilbert Syndrome).
  2. Creatinine levels: >2 mg/dL (>177 μmol/L)
* The participant is refractory to prior PPI therapy as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants at Week 12 Achieving Peak Esophageal Intraepithelial Eosinophil Count <15 eos/hpf. | Week 12

SECONDARY OUTCOMES:
Mean Change from Baseline to Week 12 in Dysphagia Days | Baseline and Week 12
Mean Change from Baseline to Week 12 in EoE Endoscopic Reference Score (EREFS). | Baseline and Week 12
Mean Change from Baseline to Week 12 in Peak Esophageal Intraepithelial Eosinophil Count. | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (36):
- United States (36):
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - GW Research, Inc, Chula Vista, California
  - Southern California Research Institute Medical Group, Los Angeles, California
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Nature Coast Clinical Research, Inverness, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - International Center for Research, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Grand Teton Research Group, Idaho Falls, Idaho
  - GI Alliance - Gurnee, Gurnee, Illinois
  - Combined Gastro, LLC, Lafayette, Louisiana
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Boston Specialists, Boston, Massachusetts
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Advanced Research Institute, Reno, Nevada
  - GCGA Physicians, LLC dba/Gastro Health Research, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research LLC, Mentor, Ohio
  - Galen Medical Group - Galen Digestive Health, Chattanooga, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - GI Alliance, Cedar Park, Texas
  - The Hospitals of Providence Memorial Campus, El Paso, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - Houston Endoscopy and Research Center, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Pearland Physicians, Pearland, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Texas Gastro Consultants, Tomball, Texas
  - Care Access - Ogdon, Ogden, Utah
  - Advanced Research Institute, Ogden, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No